CLINICAL TRIAL: NCT06905457
Title: Comparative Effect of Vojta Therapy and Bobath Therapy on Lower Limb Spasticity and Motorcity Among Hemiparetic Stroke Patients
Brief Title: Comparative Effect of Vojta Therapy and Bobath Therapy on Lower Limb Spasticity and Motorcity Among HS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/786
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vojta therapy (Experimental)
  Interventions: Combination Product: Vojta therapy
- Bobath therapy (Experimental)
  Interventions: Combination Product: Bobath therapy

INTERVENTIONS:
Combination Product: Vojta therapy — Vojta therapy, also known as Reflex Locomotion Therapy, is a specialized physiotherapy technique developed by Czech neurologist Václav Vojta, using sensory stimulation to activate innate movement patterns and improve motor skills, posture, and overall function
  Arms: Vojta therapy
Combination Product: Bobath therapy — Bobath therapy, also known as Neurodevelopmental Treatment (NDT), is a problem-solving approach to neurological rehabilitation, focusing on motor learning and efficient motor control to improve function and participation in daily activities
  Arms: Bobath therapy

SUMMARY:
Background: Stroke is clinical defined as a neurological syndrome characterized by acute disruption of blood flow to an area of brain and corresponding onset of neurological defects related to the concerned area of brain. Hemiplegic patient primarily affects the upper limb and lower limb of one side and typically results in flaccidity and difficulties with motor control and function.

DETAILED DESCRIPTION:
The aim of this study will compare the Effect of Vojta therapy and Bobath therapy on lower limb spasticity and motorcity among hemiparetic stroke patients. Methodology: Randomize clinical trials will be carried out on lower limb spasticity and motorcity among hemiparetic stroke patients. This study will include adult's stroke (1-4 months post- onset). Inclusion criteria in which diagnosed with hemiplegic patients, aged 25-75 years and willingness to participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hemiparetic stroke.
* adult's stroke (1-4 months post- onset)
* Ability to follow instructions and participate in testing
* Aged 25-75 years.

Exclusion Criteria:

* Previous history of brain surgery.
* Pregnant women.
* Limitation in cognitive skills like Aphasia, deteriorated consciousness or dementia.
* Severe cardiovascular disease (unstable hypertension)"

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment scale(FMA) | 12 Months
  The total possible scale score is 226. Points are divided among the domains as follows: Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
Modified ashworth scale( MAS) | 12 Months
  The Modified Ashworth Scale (MAS) is a clinical tool used to measure spasticity, a velocity-dependent increase in muscle stretch reflexes, by assessing the resistance to passive movement. It's a six-level ordinal scale, ranging from 0 (no increase in tone) to 4 (affected part rigid)

CONTACTS AND LOCATIONS:
Locations (1):
- Aqsa physiotherapy clinic, Main Sheikhupura road near Sitara Velly, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No